CLINICAL TRIAL: NCT04278872
Title: A Phase 2, Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of SJX-653 in Postmenopausal Women With Moderate to Severe Vasomotor Symptoms
Brief Title: Phase 2 Study of SJX-653 in Postmenopausal Women With Moderate to Severe Vasomotor Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early as the goal of determining a safe and efficacious dose for further development for the treatment of VMS was not met
Sponsor: Sojournix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJX-653-006
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — SJX-653

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SJX-653 (Experimental): Participants will receive SJX-653
  Interventions: Drug: SJX-653
- Placebo (Placebo Comparator): Participants will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SJX-653 — administered orally once daily
  Arms: SJX-653
Drug: Placebo — administered orally once daily
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy, safety, tolerability, and pharmacokinetics of once daily SJX-653 in postmenopausal women with moderate to severe VMS.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a consent form before Screening procedures begin.
2. Be a postmenopausal female, 40 to 65 years of age (inclusive) at the Screening Visit, defined as:

   1. Spontaneous amenorrhea for at least 12 months, OR
   2. 6 months of spontaneous amenorrhea with serum FSH levels >40 milli-International unit (mIU/mL), OR
   3. 6 weeks past a postsurgical bilateral oophorectomy with or without hysterectomy.

   All postmenopausal woman (PMW) must have a serum follicle stimulating hormone (FSH) >40 mIU/mL at Screening.
3. Have an average of at least 7 moderate to severe VMS per day at Baseline. The following definitions for severity are used:

   1. Mild: Sensation of heat without sweating/damping; if at night, do not wake up but later notice damp sheets or clothing.
   2. Moderate: Sensation of heat with sweating/dampness, but able to continue activity; if at night, wake up because hot and/or sweating, but no action is necessary other than rearranging the bed sheets.
   3. Severe: Sensation of heat with sweating causing disruption of current activity; if at night, wake up hot and sweating and need to take action (eg, removing layer of clothes, open the window, or get out of bed).
4. Have a body mass index between 18 and 35 kg/m2, inclusive.
5. For subjects 50-65 years old, have documentation (written or electronic report) of a satisfactory mammogram result at Screening within applicable intervals stated in local breast cancer screening guidelines. Subjects 40-49 years old require a mammogram within the same intervals.
6. Have documentation (written or electronic report) of a normal Pap smear (or equivalent cervical cytology) ) in combination with Human Papilloma virus (HPV) testing, or a Pap smear of no clinical significance in the opinion of the Investigator, at Screening within applicable intervals stated in local cervical cancer prevention guidelines.
7. Have an endometrial thickness ≤4 mm by transvaginal ultrasound at Screening.
8. Be willing to undergo an endometrial biopsy if they have unexplained bleeding during the study or endometrial thickness >4 mm at the EOT visit. An endometrial biopsy is not required for subjects who have had a partial (supracervical) or full hysterectomy.

Exclusion Criteria:

1. Have clinically significant history or evidence of poorly controlled cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s) as determined by the Investigator or have any medical condition that requires chronic medication and that in the Investigator's opinion, would make subjects unsuitable for participation in the study.
2. Have manifest or suspected active COVID-19 infection. Have tested positive for presence of SARS-CoV-2 based on a RT-PCR or other validated test; or have clinical symptoms suggestive of COVID-19 infection; or have to comply with quarantine requirements per local Public Health directive.
3. Have a history of diagnosis of major depressive disorder in the 3 years prior to Screening, or are on any antidepressant, anxiolytic or antipsychotic treatment. Selective serotonin reuptake inhibitors (SSRIs) and serotonin and norepinephrine reuptake inhibitors (SNRIs) treatment for mild depression and/or mild anxiety is allowed provided medication is stable and well-tolerated in the 3 months prior to the Screening Visit and does not change during study participation.
4. Have a history of suicide ideation or attempt in the past 3 years.
5. Have a history of a sleep disorder other than insomnia due to VMS (eg, narcolepsy, sleep apnea, restless leg syndrome).
6. Have clinical or biochemical evidence of active hepatitis or other significant hepatic or biliary disease (eg, chronic hepatitis, cirrhosis, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, nonalcoholic steatohepatitis, nonalcoholic fatty liver disease, or hereditary liver disease).
7. Have any abnormal liver function tests at Screening or an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (CKD-EPI 2009 calculation; Levey et al 2009).
8. Have tested positive for human immunodeficiency virus, hepatitis B, C or E at Screening.
9. Have any gastrointestinal, liver, kidney or other disorder that would significantly interfere with the absorption, distribution, metabolism, or excretion (ADME) of drugs in the opinion of the Investigator.
10. Have a history of alcohol abuse or a history of substance abuse.
11. Smoking >10 cigarettes per day.
12. Regularly working night shifts.
13. Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg, based on the median of a total of 4 to 6 readings, from 2 to 3 readings taken on 2 diﬀerent occasions.
14. Have clinically significant abnormal ECG or QT interval prolongation (corrected for heart rate using Fridericia formula [QTcF] prolongation >470 ms) at Screening.
15. Have a history of endometrial hyperplasia or uterine/endometrial cancer.
16. Have current unexplained uterine bleeding.
17. Have a history of cancer prior to Screening (other than local, treated basal cell or squamous cell carcinoma).
18. Have any significant illness requiring hospitalization or emergency treatment within 4 weeks prior to the Screening Visit or during the Screening or Run-in Periods, and as determined by the Investigator.
19. Are pregnant or lactating.
20. Have used hormonal treatments within defined periods of time prior to the start of the Run-in Period. Washout times dependent on treatment.
21. Are taking any nonhormonal medication for treatment of VMS in the 8-week period prior to the start of the Run-in Period.
22. Have used herbal supplements or over-the-counter (OTC) medications for treatment of VMS 8 weeks prior to the start of the Run in Period. Any other herbal supplements or OTC supplements that could interfere with the study objectives require a 28-day wash-out period prior to the start of the Run-in Period.
23. Are taking any antiestrogens, selective estrogen receptor modulators, or aromatase inhibitors.
24. Are taking any antigonadotropin medication.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sojournix, Inc.
Locations (22):
- Belgium (3):
  - Sojournix Site #202, Brussels
  - Sojournix Site #204, Genk
  - Sojournix Site #201, Ghent
- Germany (6):
  - Sojournix Site #308, Berlin
  - Sojournix Site #309, Berlin
  - Sojournix Site #304, Bernburg
  - Sojournix Site #301, Hamburg
  - Sojournix Site #306, Hamburg
  - Sojournix Site #305, Marburg
- Poland (6):
  - Sojournix Site #401, Bialystok
  - Sojournix Site #402, Katowice
  - Sojournix Site #406, Lodz
  - Sojournix Site #403, Lublin
  - Sojournix Site #404, Lublin
  - Sojournix Site #405, Lublin
- United Kingdom (7):
  - Sojournix Site #108, Blackpool
  - Sojournix Site #111, Cannock
  - Sojournix Site #104, Glasgow
  - Sojournix Site #112, Leeds
  - Sojournix Site #110, Liverpool
  - Sojournix Site #105, London
  - Sojournix Site #107, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SJX-653 | Placebo
Started | 7 | 6
Completed | 4 | 5
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Study Termination | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SJX-653 | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (3.29) | 58.3 (4.03) | 57.2 (3.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Average Daily Frequency of Moderate to Severe Vasomotor Symptoms (VMS) From Baseline to Week 4
Description: Moderate to severe vasomotor symptoms collected daily by e-diary
Time Frame: Baseline to Week 4
Population: Study was terminated early and program discontinued. Raw data (patient-reported outcomes/diary entries) were not processed to obtain primary outcome measures, therefore primary outcome measures could not be analyzed.
Arm/Group | SJX-653 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Change in the Severity of Moderate to Severe VMS From Baseline to Week 4
Time Frame: Baseline to Week 4
Reporting Status: Not Posted

3. Secondary Outcome: Mean Change and Percent Change of Parameters of VMS Frequency and Severity by Study Week
Time Frame: Baseline up to Week 6
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change From Baseline in Insomnia Severity Index (ISI)
Time Frame: Baseline up to Week 4
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change From Baseline in Hot Flash Related Daily Interference Scale (HFRDIS)
Time Frame: Baseline up to Week 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Treatment-Emergent Adverse Events
Arm/Group | SJX-653 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/7 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJX-653 (N=7) | Placebo (N=6)
Constipation (Gastrointestinal disorders) | 1 (3) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
LDH increased (Investigations) | 1 (1) | 0 (0)
GLDH increased (Investigations) | 1 (1) | 0 (0)
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
SARS-Cov-2 test positive (Investigations) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04278872/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT04278872/SAP_001.pdf